CLINICAL TRIAL: NCT02180503
Title: Relative Bioavailability of 1 mg and 10 mg BI 1356 BS as Powder in the Bottle (PIB) Reconstituted With 0.1% Tartaric Acid Compared to 1 mg and 10 mg BI 1356 BS as Tablets as Single Oral Administration in Healthy Male Volunteers (Separately at Each Dose Level) Including the Influence of Food (Standardised High Fat Breakfast) on the Bioavailability of 10 mg BI 1356 BS as Tablet in a Single Dose, Open-label, Randomised, Two-way (1 mg) and Three-way (10 mg) Crossover Trial
Brief Title: Relative Bioavailability of 1 mg and 10 mg BI 1356 BS as Powder in the Bottle (PIB) to 1 mg and 10 mg BI 1356 BS as Tablets as Single Oral Administration in Healthy Male Volunteers Including the Influence of Food on the Bioavailability of 10 mg BI 1356 BS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.8
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Food

ARMS (2):
- BI 1356 BS - low dose (Experimental)
  Interventions: Drug: BI 1356 BS PIB - low dose; Drug: BI 1356 BS tablet - low dose
- BI 1356 BS - high dose (Experimental)
  Interventions: Drug: BI 1356 BS PIB - high dose; Drug: BI 1356 BS tablet - high dose; Drug: BI 1356 BS tablet - high dose with food

INTERVENTIONS:
Drug: BI 1356 BS PIB - low dose
  Arms: BI 1356 BS - low dose
Drug: BI 1356 BS tablet - low dose
  Arms: BI 1356 BS - low dose
Drug: BI 1356 BS PIB - high dose
  Arms: BI 1356 BS - high dose
Drug: BI 1356 BS tablet - high dose
  Arms: BI 1356 BS - high dose
Drug: BI 1356 BS tablet - high dose with food
  Arms: BI 1356 BS - high dose

SUMMARY:
Investigation of the relative bioavailability of 1 mg and 10 mg BI 1356 BS as PIB reconstituted with 0.1% tartaric acid vs. 1 mg and 10 mg BI 1356 BS as tablet including a food effect for the 10 mg tablet dose group

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP),Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests

  * No findings deviating from normal and of clinical relevance
  * No evidence of a clinically relevant concomitant disease
* Age ≥21 and Age ≤65 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* No adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until one month after the last intake

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-08; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | Up to 264 h after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | Up to 264 h after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 264 h after drug administration
AUCt1-t2 (Partial area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) | Up to 264 h after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | Up to 264 h after drug administration
λz (terminal rate constant in plasma) | Up to 264 h after drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 264 h after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | Up to 264 h after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Up to 264 h after drug administration
Number of patients with adverse events | Up to 18 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | Up to 18 days after last drug administration
Clinically relevant changes in clinical laboratory values | Up to 18 days after last drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | Up to 264 h after drug administration